CLINICAL TRIAL: NCT05496361
Title: A Prospective, Multi-center and Randomized Controlled Clinical Trial to Assess the Safety and Effectiveness of Tianyi Revascularization Device of in the Revascularization of Large Vessel Occlusion in Acute Ischemic Stroke
Brief Title: A Prospective, Multi-center and Randomized Controlled Trial of Tianyi Revascularization Device in Acute Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Zenith Vascular Scitech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTP-301
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: AIS; Acute Ischemic Stroke; Large Vessel Occlusion; Thrombectomy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tianyi Revascularization Device (Experimental)
  Interventions: Device: Tianyi Revascularization Device
- Solitaire FR Revascularization Device (Active Comparator)
  Interventions: Device: Solitaire FR Revascularization Device

INTERVENTIONS:
Device: Tianyi Revascularization Device — Revascularization Device using the Mechanical thrombectomy technique for recanalization of an occlusion large vessel in the brain
  Arms: Tianyi Revascularization Device
Device: Solitaire FR Revascularization Device — Revascularization Device using the Mechanical thrombectomy technique for recanalization of an occlusion large vessel in the brain
  Arms: Solitaire FR Revascularization Device

SUMMARY:
This is a prospective, randomized, single blind, concurrent controlled, multi-center study. Patients presenting with symptoms of acute ischemic stroke who have evidence of a large vessel occlusion in the cerebral circulation.

DETAILED DESCRIPTION:
This is a prospective, randomized, single blind, concurrent controlled, multi-center study. Patients presenting with symptoms of acute ischemic stroke who have evidence of a large vessel occlusion in the cerebral circulation will be assigned to either the Tianyi Revascularization Device or Solitaire FR Revascularization Device. Each treated patient will be followed and assessed for 3 months after randomization. Up to 238 evaluable patients at up to 18 centers presenting with acute ischemic stroke in vessels accessible to the Revascularization Device for revascularization within 8 hours of symptom onset. The hypothesis to be tested is that the safety and effectiveness of the Tianyi Revascularization Device for the revascularization of large vessel occlusion is not inferior to the Solitaire FR Revascularization Device.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-85 years
2. within 8 hours after symptom onset
3. The results showed that the scores of ASPECTS ≥6, 0<NIHSS<30 , and mRS <2 ;
4. caused by a large vessel occlusion of the anterior circulation (internal carotid artery or the M1 and M2 segments of MCA and the A1 and A2 segments) cerebral artery confirmed by DSA;
5. Signed informed consent.

Exclusion Criteria:

Clinical exclusion criteria:

1. Patients with epileptic seizure during stroke;
2. Patients with life expectancy less than 90 days;
3. Patients with intracranial hemorrhage or subarachnoid hemorrhage on the same side in recent 3 months;
4. Previous history of intracranial tumor, cerebral arteriovenous malformation or aneurysm without surgical treatment
5. Patients with a history of cerebral infarction or myocardial infarction or uncontrolled serious infectious diseases (such as endocarditis or septicemia) in recent 3 months;
6. Patients with gastrointestinal or urinary tract bleeding in the past three weeks;
7. Patients who have participated in clinical trials of other drugs or devices and have not been withdrawn from the group within the first one months of the screening period of this trial;
8. Patients with serious mental history, heart, liver, lung and kidney failure or other serious diseases;
9. Patients with active bleeding or known bleeding tendency (INR>3.0 or platelet count<40*10^9/L or APTT>50 seconds);
10. The blood glucose which could not be controlled by drugs was less than 2.7 mmol/L or more than 22.2 mmol/L;
11. Patients with hypertension beyond the control of drugs (systolic blood pressure >180 mmHg, or diastolic blood pressure >105 mmHg);
12. Females who are pregnant or in lactation;
13. Patients who are known to be allergic or resistant to contrast agents, anesthetics, anticoagulants, antiplatelet drugs and nickel-titanium;
14. Patients who have undergone major surgical operations in the past month;
15. Other cases with unknown onset time or unsuitable for inclusion in the group judged by researchers;other conditions not suitable for inclusion judged by the researcher;

Imaging exclusion criteria

1. Patients with intracerebral hemorrhage confirmed by CT (except for microbleeds. At the discretion of each Investigator);
2. ASPECTS <6 points on head CT;
3. Patients with common carotid artery occlusion who are known or suspected to be chronic occlusion;
4. DSA showed that bilateral carotid system was occluded at the same time;
5. DSA showed (or highly suspected) carotid dissection or arteritis;
6. DSA showed that the vascular route was tortuous, and the device was difficult to reach the target position or recover;
7. Subjects who are not eligible for inclusion after imaging review in the group judged by researchers.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2021-01-24 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Revascularization assessed by digital subtraction angiography of the occluded target vessel to mTICI 2b or 3 at immediate post-procedure | At immediate post-procedure

SECONDARY OUTCOMES:
Times to revascularization（From groin puncture to final revascularization result） | At immediate post-procedure
NIHSS score at 24h, 7-day or discharge | Within 24 hours，7-day or discharge post-procedure, whichever came first
Functional patient outcome at 90 days post-procedure as defined by a modified Rankin Score (mRS) 0-2 | at 90 days post-procedure
Device Technical Success | At immediate post-procedure

OTHER OUTCOMES:
Occurrence of symptomatic intracranial hemorrhages (sICH) at 24 hours | Within 24 hours post-procedure
All causes of mortality at 90 days | at 90 days post-procedure
Occurrence of serious adverse events or adverse events related to device or procedure | at 90 days post-procedure
Occurrence of device defect | at 90 days post-procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No